CLINICAL TRIAL: NCT06039540
Title: A Comprehensive Research of Pediatric Heart Failure--A Prospective Cohort Study of Drug Therapy for Pediatric Heart Failure
Brief Title: Study of Drug Therapy for Pediatric Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Peking University First Hospital (Other); Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Shoujun Li, Director of Congenital Heart Surgery Center, China National Center for Cardiovascular Diseases
Other Study IDs: 2022-1-4032-1
Record Dates: First submitted 2023-09-09; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Heart Failure Congenital
Keywords: congenital heart failure; drug therapy; congenital heart disease postoperative
MeSH Terms: interventions — Captopril; Metoprolol; Spironolactone; Torsemide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Modified Drug Therapy Group: Patient in this group will undergo a one-year course of medication, including Captopril(tablet, 0.3mg/kg, tid), Metoprolol(tablet, 0.2mg/kg, bid), Spironolactone(tablet, 2-4mg/kg, bid), Torsemide(tablet, 0.2-0.5mg/ mg, bid), and Potassium Citrate(powder, 0.06g/kg, tid).e Traditional Drug Therapy Group
  Interventions: Drug: Captopril Tablets; Drug: Metoprolol Oral Tablet; Drug: Spironolactone Tablets; Drug: Torsemide Tablets; Drug: Potassium citrate powder
- Traditional Drug Therapy Group: Patient in this group will undergo a one-year course of medication, including Torsemide(tablet, 0.2-0.5mg/mg, bid) and Potassium Citrate(powder, 0.06g/kg, tid).
  Interventions: Drug: Torsemide Tablets; Drug: Potassium citrate powder

INTERVENTIONS:
Drug: Captopril Tablets — 0.3mg/kg, tid
  Groups: Modified Drug Therapy Group
Drug: Metoprolol Oral Tablet — 0.2mg/kg, bid
  Groups: Modified Drug Therapy Group
Drug: Spironolactone Tablets — 2-4mg/kg, bid
  Groups: Modified Drug Therapy Group
Drug: Torsemide Tablets — 0.2-0.5mg/mg, bid
Drug: Potassium citrate powder — 0.06g/kg, tid

SUMMARY:
The goal of this observational study is to compare the safety and effectiveness of a modified drug therapy with traditional drug therapy in pediatric heart failure patients.

The main questions it aims to answer are:

* Can a modified drug therapy improve left ventricular function in pediatric heart failure patients?
* Can the adverse drug reactions caused by the modified drug therapy be non-inferior (clinically acceptable) to those of the traditional drug therapy? Participants will be assigned to either the Modified Drug Therapy Group (comprising angiotensin-converting enzyme inhibitor (ACE-I), beta-blockers, diuretics, potassium supplements, and spironolactone) or the Traditional Drug Therapy Group (diuretics and potassium supplements) based on personal preferences and clinical assessments by their attending physicians. They will undergo a 6-months course of medication. Additionally, echocardiography, electrocardiograms, complete blood counts, biochemical tests, and measurements of N-terminal pro-brain natriuretic peptide (NT-proBNP) were conducted before the initiation of medication therapy and at 1 month, 3 months, and 6 months after treatment commencement. Researchers will compare the Modified Drug Therapy Group and the Traditional Drug Therapy Group to see if the recurrence rate of moderate to severe mitral valve regurgitation, as assessed by echocardiography after 6 months of treatment, is lower in the former than in the latter.

ELIGIBILITY:
Inclusion Criteria:

* Patients younger than 14 years of age
* heart failure after congenital heart surgery
* Ross > 2 or NYHA > 2
* LVEF<55%, or LVFS<25%

Exclusion Criteria:

* single ventricle
* congenital heart disease without anatomical correction
* Patients with heart failure requiring ventricular assist or cardiac synchronization therapy
* Patients with severe pulmonary hypertension (pulmonary arterial pressure >6 Wood·U)
* Patients with severe liver and kidney failure
* Patients who are allergic to related medications
* Patients with symptomatic hypotension who cannot tolerate related drugs
* Refuse to sign the informed consent or refuse to participate in this experiment

Max Age: 14 Years | Sex: All
Age Groups: Child
Study Population: paitent younger than 14 years of age with heart failure after suergry congenital heart disease
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-06-22 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the recurrence rate of heart failure | after 6 months of treatment
  During follow-up visits, echocardiographic examination is conducted to measure the left ventricular function. If LVEF falls under 55%, it is recorded as a recurrence.

SECONDARY OUTCOMES:
NT-proBNP level | after 6 months of treatment
  The trend in NT-proBNP levels.
Incidence rate of drug adverse reactions | after 6 months of treatment
  The incidence of abnormalities in complete blood count, electrolytes, liver and kidney function, and cardiac enzymes.
Readmission rate for heart failure | after 6 months of treatment
  During follow-up visits, readmission for heart failure will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Shoujun Li, MD, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No